CLINICAL TRIAL: NCT03883529
Title: Reviewing Birth Experience With a Known Midwife: a Feasibility Study
Brief Title: Reviewing Birth Experience With a Known Midwife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIceland
Record Dates: First submitted 2019-02-21; First posted 2019-03-21 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Childbirth
Keywords: Birth experience; Midwifery; Feasibilty; Intervention

STUDY DESIGN:
Intervention Model Description: The study is a pilot feasibility study, exploring a new type of intervention after birth, for women who had their antenatal care provided at a high-risk maternity clinic. The intervention involves women writing about and reviewing their birth experience, six to eight weeks after birth, with the midwife who provided antenatal care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women reviewing birth experience (Experimental): Women who had their antenatal care provided at a high-risk antenatal clinic, will be offered to write about and review their birth experience about 6 weeks post-partum with a known midwife from antenatal care.
  Interventions: Other: Writing about and reviewing birth experience

INTERVENTIONS:
Other: Writing about and reviewing birth experience — Writing about and reviewing birth experience with a known midwife from antenatal care about 6 weeks post-partum.

SUMMARY:
The study is a part of a PhD thesis. The study aims to develop a specific midwifery intervention consisting of two components; women writing about the birth experience and reviewing their experience with a known midwife. Women´s birth experience has received research attention worldwide, showing a prevalence of negative birth experience ranging from 5-34%. Considerable knowledge of predictors and impacts of negative birth experience exists, but less is known about effective interventions although women report that reviewing birth experiences is beneficial. Six to eight midwives, providing antenatal care at the high-risk maternity clinic at Landspitali University Hospital, provide the intervention after completing a special training program. Thirty women who had their antenatal care provided at the clinic, after 28 weeks of pregnancy, will be invited to write about their birth experience and review it with the midwife who provided their antenatal care, four to six weeks after birth. The study is based on a mixed method design where quantitative and qualitative data will be collected. Data including traumatic symptoms, birth outcomes, birth experience and experience of the intervention, will be collected from women before the intervention and then six weeks later. The participating midwives´ diaries and focus group interviews will be used to explore their experience of providing the intervention. Descriptive and thematic analysis will be used.

DETAILED DESCRIPTION:
The purpose of the study is to develop and explore the feasibility and acceptability of an intervention, involving writing about and reviewing birth experience with a known midwife from antenatal care.

Studies in developed countries indicate that between 5-16.5% of women perceive their births to be negative. The perception of birth experience seems to be consistent over time, suggesting that time alone does not have a healing effect. Adverse consequences of negative birth experience can be profound and have an impact on different aspects of woman´s life. Among well-known consequences are development of fear of childbirth, a tendency to delay pregnancy and longer interval between children, an increase in request for elective caesarean section without health indications and mental health problems like depression, anxiety and post-traumatic stress disorder (PTSD). Around 1-6% of women develop PTSD in response to pregnancy, birth and post-partum events. Negative birth experience may have long-term and negative consequences on the women´s self-identity and relationships with their infants and partners. This is of concern as there is a growing body of literature showing negative consequences of maternal mental distress on the mother-infant bonding and attachment process, and relationships with partner. Improvement in bonding could take as long as one to five years - which needs attention because a delay in bonding can have detrimental effects on the child's long-term development.

Risk factors for a negative birth experience are multifaceted and associations have been found between negative birth experience and instrumental or caesarean births, intrapartum complications, maternal complications or hospitalisation in pregnancy and prolonged labour. Furthermore, fear of childbirth, negative thoughts about the upcoming birth, prior negative birth experience, feelings of not being in control, and powerlessness during birth have been associated with negative birth experiences as well as history of mental health problems. Furthermore, perceived lack of professional support during pregnancy or birth has been associated with negative experience of birth.

Evidence for useful methods to assist women with negative childbirth experience is limited. Interventions aimed to assist women with negative birth experience have been explored but the effectiveness remains inconsistent, with five comparative studies showing improvements on psychological measures while six of them did not. In recent studies a method of writing about the experience was explored with promising results, where one of them showed a reduction in depressive and traumatic symptoms and the other one showed emotional benefits like clarifying thoughts and feelings of empowerment.

It is worth considering that in many of the above comparative studies, the need to review the birth experience was based on the view of health professionals. Also, the interviews were limited to women who experienced an operative birth or unexpected events during birth but none of these were effective in psychological improvements. Likewise, the time between the negative birth experience until the intervention was provided ranged from the first week after birth up to seven years after birth. Similarly, the structure, content and quantity of interview interventions varied. Each study´s design and outcome measures used, varied significantly making it difficult to determine which components of the interventions women considered most effective. Despite failure in these studies to show significant changes in psychological measures, women reported that it was helpful to participate in the intervention.

The results from authors´ recent study in Iceland provide important insights into women´s views about the process of reviewing negative birth experience and reconciling difficult emotions, at a special midwifery clinic Ljáðu mér eyra (LME) at Landspítali. The women prefer their negative birth experiences to be detected by professionals and consequently have opportunity to review their birth experience in a tailored conversation on their terms. Many of them revealed preferences of talking to a known midwife who had provided care during pregnancy or birth, suggesting a request for some form of continuity of care. Reviewing the birth experience provided an opportunity for many women to relieve the burden of difficult emotions, enhance well-being and gain strength to move on with their lives.

The ideological background of the study is affected by the international ideology of midwifery and models of care. According to the International Confederation of midwives' philosophy and model of midwifery care (2014), birth is not only … a normal and physiological process… but also … a profound experience, which carries significant meaning to the woman and her family. Midwifery care combines art and science and is holistic in nature, grounded in an understanding of the social, emotional, cultural, spiritual, psychological experiences of women and based upon the best available evidence. Furthermore, in International Confederation of midwives' code of ethics (2014) is stated that midwives should … respond to the psychological, physical, emotional and spiritual needs of women…,requiring midwives to react to women´s needs following childbirth from a holistic perspective. This philosophy of care is extended in Renfrew´s et. al. framework for childbirth care and a midwifery model of woman-centred childbirth care, developed in Swedish and Icelandic settings. Good quality midwifery care includes continuity of care, information, communication and understanding of women's needs. According to the above, interventions need to be tailored to women's circumstances and needs and provided in partnership with them.

Thirty women who had their antenatal care provided at the clinic, after 28 weeks of pregnancy, will be invited to write about their birth experience and review it with the midwife who provided their antenatal care, four to six weeks after birth. Six to eight midwives will provide the intervention after completing a 12-hour training program. The study is based on a mixed method design where quantitative and qualitative data will be collected. Data including traumatic symptoms, traumatic life events, birth outcomes and birth experience will be collected from women before the intervention. Four to six weeks after the intervention, data about birth experience, traumatic symptoms and experience of the intervention will be collected. The participating midwives´ diaries and focus group interviews will be used to explore their experience of providing the intervention. Descriptive and thematic analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years old, having their antenatal care provided at the clinic after 28 weeks of pregnancy and planned a vaginal birth.

Exclusion Criteria:

* Women < 18 years old, referred to the clinic after 28 weeks of pregnancy, not reading Icelandic or planned elective caesarean section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in traumatic symptoms | 4-6 weeks and 10-12 weeks post-partum
  The Icelandic version of the Post-traumatic stress disorder Checklist for DSM-5 (PCL-5) will be used. It is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of post-traumatic stress disorder. The self-reporting rating scale is 0-4, from ´Not at all,´ ´A little bit,´ Moderately,´ ´Quite a bit,´ to ´Extremely´. A total symptom severity score ranges from 0-80, with higher scores indicating more post-traumatic symptoms. It can also be interpreted in clusters of avoidance (5 items), avoidance (2 items), negative alterations in cognitions and mood (7 items) and alterations in arousal and reactivity (6 items).
Traumatic events in lifetime | 4-6 weeks
  Traumatic events in lifetime are measured with the Life Events Checklist for DSM-5 (LEC-5), translated in Icelandic. The LEC-5 is a self-report measure to screen for potentially traumatic events in a respondent's lifetime. It assesses exposure to 16 events known to potentially result in traumatic symptoms and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale: ´happened to me´, ´witnessed it´, ´learned about it´, ´part of my job´, ´not sure´, ´doesn't apply´.
Change in the perception of birth experience | 4-6 weeks and 10-12 weeks post-partum
  The birth experience will be measured by responses from the question ´How did you experience your birth?´ with the response options ranging from 1 (very positive) to 5 (very negative)
Change in the overall perception of birth experience | 4-6 weeks and 10-12 weeks post-partum
  The birth experience will be measured by responses from the question ´How was your overall perception of your birth?´ with the response options ranging from 1 (very difficult) to 5 (very easy).
Self-reported birth outcomes: onset of labour, birth mode, experience of the birth duration, admission to neonatal intensive care unit, perineal outcomes and breastfeeding | 4-6 weeks post-partum
  Information about birth outcomes will be obtained by questions about the onset of labour, birth mode, experience of the birth duration, admission to neonatal intensive care unit and perineal outcomes. Breastfeeding will be addressed by the question ´How did you perceive the breastfeeding was going?´ with options on a five-point Likert scale 1 (very well) to 5 (very bad) or ´I did not breastfeed'.
Change in self-reported well-being during recent birth | 4-6 weeks and 10-12 weeks post-partum
  Information about well-being during the recent birth will be obtained by a list of statements f.ex. ´I felt secure/strong/in control´ with response options ranging from 1 (very much agree) to 5 (very much disagree)
Self-reported health-related issues before and during pregnancy | 4-6 weeks post-partum
  Information about health-related issues will be obtained by a list of common health problems known to increase risk during the childbirth period. The list includes statements of physical or mental health issues f.ex. 'I have a history of or had diabetes/hypertension/mental disorders... before pregnancy', with the option ´other´ at the end (free text). Health during the recent pregnancy will be obtained by a list of common risk factors during pregnancy f.ex. ´I was diagnosed with diabetes/hypertension/pre-eclampsia/... during pregnancy´, with the option ´other´ (free text) at the end.
Self-reported reproductive history | 4-6 weeks post-partum
  Information about reproductive history will be obtained by a list of statements about parity and history of premature birth, stillbirth, placenta abruptio, emergency cesarean or fear of birth.
Perception of writing about and reviewing birth experience with a known midwife | 10-12 weeks post-partum
  Women´s perception of reviewing the birth experience will be obtained by questions about if the intervention; was useful, met their expectations, they got answers to their questions, if they felt they were listened to and could express themselves. The responses were on a five-point Likert scale from 1 (very much agree) to 5 (very much disagree). They will also be asked of their views about the conversation about reviewing the birth experience, when, where and who should provide it. Space for free text reports about the interview will be at the end of the questionnaire.
Socio-demographic factors: age, education, marital status, | 4-6 weeks post-partum
  The age will be measured by year of birth. The educational status and marital status will be measured by lists of four categories.

CONTACTS AND LOCATIONS:
Overall Officials: Helga Gottfredsdottir, Study Director — University of Iceland
Locations (1):
- Valgerdur Lisa Sigurdardottir, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigurdardottir VL, Gamble J, Gudmundsdottir B, Kristjansdottir H, Sveinsdottir H, Gottfredsdottir H. The predictive role of support in the birth experience: A longitudinal cohort study. Women Birth. 2017 Dec;30(6):450-459. doi: 10.1016/j.wombi.2017.04.003. Epub 2017 May 3. PMID 28478933
- [Background] Sigurethardottir VL, Gamble J, Guethmundsdottir B, Sveinsdottir H, Gottfreethsdottir H. Processing birth experiences: A content analysis of women's preferences. Midwifery. 2019 Feb;69:29-38. doi: 10.1016/j.midw.2018.10.016. Epub 2018 Oct 27. PMID 30396158
- [Background] Rijnders M, Baston H, Schonbeck Y, van der Pal K, Prins M, Green J, Buitendijk S. Perinatal factors related to negative or positive recall of birth experience in women 3 years postpartum in the Netherlands. Birth. 2008 Jun;35(2):107-16. doi: 10.1111/j.1523-536X.2008.00223.x. PMID 18507581
- [Background] Waldenstrom U, Hildingsson I, Rubertsson C, Radestad I. A negative birth experience: prevalence and risk factors in a national sample. Birth. 2004 Mar;31(1):17-27. doi: 10.1111/j.0730-7659.2004.0270.x. PMID 15015989
- [Background] Ayers S, Eagle A, Waring H. The effects of childbirth-related post-traumatic stress disorder on women and their relationships: a qualitative study. Psychol Health Med. 2006 Nov;11(4):389-98. doi: 10.1080/13548500600708409. PMID 17129916
- [Background] Fenech G, Thomson G. Tormented by ghosts from their past': a meta-synthesis to explore the psychosocial implications of a traumatic birth on maternal well-being. Midwifery. 2014 Feb;30(2):185-93. doi: 10.1016/j.midw.2013.12.004. Epub 2013 Dec 13. PMID 24411664
- [Background] Waldenstrom U. Why do some women change their opinion about childbirth over time? Birth. 2004 Jun;31(2):102-7. doi: 10.1111/j.0730-7659.2004.00287.x. PMID 15153129
- [Background] Baxter JD, McCourt C, Jarrett PM. What is current practice in offering debriefing services to post partum women and what are the perceptions of women in accessing these services: a critical review of the literature. Midwifery. 2014 Feb;30(2):194-219. doi: 10.1016/j.midw.2013.12.013. Epub 2013 Dec 27. PMID 24491690
- [Background] Borg Cunen N, McNeill J, Murray K. A systematic review of midwife-led interventions to address post partum post-traumatic stress. Midwifery. 2014 Feb;30(2):170-84. doi: 10.1016/j.midw.2013.09.003. Epub 2013 Sep 21. PMID 24238899
- [Background] Gamble J, Creedy D, Moyle W, Webster J, McAllister M, Dickson P. Effectiveness of a counseling intervention after a traumatic childbirth: a randomized controlled trial. Birth. 2005 Mar;32(1):11-9. doi: 10.1111/j.0730-7659.2005.00340.x. PMID 15725200
- [Background] Lavender T, Walkinshaw SA. Can midwives reduce postpartum psychological morbidity? A randomized trial. Birth. 1998 Dec;25(4):215-9. doi: 10.1046/j.1523-536x.1998.00215.x. PMID 9892887
- [Background] Ryding EL, Wiren E, Johansson G, Ceder B, Dahlstrom AM. Group counseling for mothers after emergency cesarean section: a randomized controlled trial of intervention. Birth. 2004 Dec;31(4):247-53. doi: 10.1111/j.0730-7659.2004.00316.x. PMID 15566336
- [Background] Meades R, Pond C, Ayers S, Warren F. Postnatal debriefing: have we thrown the baby out with the bath water? Behav Res Ther. 2011 May;49(5):367-72. doi: 10.1016/j.brat.2011.03.002. Epub 2011 Mar 12. PMID 21457944
- [Background] Blasio PD, Camisasca E, Caravita SC, Ionio C, Milani L, Valtolina GG. THE EFFECTS OF EXPRESSIVE WRITING ON POSTPARTUM DEPRESSION AND POSTTRAUMATIC STRESS SYMPTOMS. Psychol Rep. 2015 Dec;117(3):856-82. doi: 10.2466/02.13.PR0.117c29z3. Epub 2015 Nov 23. PMID 26595300
- [Background] Blainey SH, Slade P. Exploring the process of writing about and sharing traumatic birth experiences online. Br J Health Psychol. 2015 May;20(2):243-60. doi: 10.1111/bjhp.12093. Epub 2014 Mar 12. PMID 24620933
- [Background] Park CL. Making sense of the meaning literature: an integrative review of meaning making and its effects on adjustment to stressful life events. Psychol Bull. 2010 Mar;136(2):257-301. doi: 10.1037/a0018301. PMID 20192563
- [Background] Bastos MH, Furuta M, Small R, McKenzie-McHarg K, Bick D. Debriefing interventions for the prevention of psychological trauma in women following childbirth. Cochrane Database Syst Rev. 2015 Apr 10;2015(4):CD007194. doi: 10.1002/14651858.CD007194.pub2. PMID 25858181
- [Background] Thomson G, Downe S. Emotions and support needs following a distressing birth: Scoping study with pregnant multigravida women in North-West England. Midwifery. 2016 Sep;40:32-9. doi: 10.1016/j.midw.2016.06.010. Epub 2016 Jun 8. PMID 27428096
- [Background] Renfrew MJ, McFadden A, Bastos MH, Campbell J, Channon AA, Cheung NF, Silva DR, Downe S, Kennedy HP, Malata A, McCormick F, Wick L, Declercq E. Midwifery and quality care: findings from a new evidence-informed framework for maternal and newborn care. Lancet. 2014 Sep 20;384(9948):1129-45. doi: 10.1016/S0140-6736(14)60789-3. Epub 2014 Jun 22. PMID 24965816
- [Background] Berg M, Asta Olafsdottir O, Lundgren I. A midwifery model of woman-centred childbirth care--in Swedish and Icelandic settings. Sex Reprod Healthc. 2012 Jun;3(2):79-87. doi: 10.1016/j.srhc.2012.03.001. Epub 2012 Mar 16. PMID 22578755
- [Background] Ferlie EB, Shortell SM. Improving the quality of health care in the United Kingdom and the United States: a framework for change. Milbank Q. 2001;79(2):281-315. doi: 10.1111/1468-0009.00206. PMID 11439467
- [Background] Turkstra E, Mihala G, Scuffham PA, Creedy DK, Gamble J, Toohill J, Fenwick J. An economic evaluation alongside a randomised controlled trial on psycho-education counselling intervention offered by midwives to address women's fear of childbirth in Australia. Sex Reprod Healthc. 2017 Mar;11:1-6. doi: 10.1016/j.srhc.2016.08.003. Epub 2016 Aug 29. PMID 28159118
- [Background] Gamble J, Creedy DK. A counselling model for postpartum women after distressing birth experiences. Midwifery. 2009 Apr;25(2):e21-30. doi: 10.1016/j.midw.2007.04.004. Epub 2007 Jul 27. PMID 17673341
- [Background] Bell AF, Rubin LH, Davis JM, Golding J, Adejumo OA, Carter CS. The birth experience and subsequent maternal caregiving attitudes and behavior: a birth cohort study. Arch Womens Ment Health. 2019 Oct;22(5):613-620. doi: 10.1007/s00737-018-0921-3. Epub 2018 Oct 23. PMID 30353272